CLINICAL TRIAL: NCT01802593
Title: Phase 4, Open Label Multicenter Randomized Controlled Trial. Comparison of 2 Immunomodulator Withdrawal Schemes for Infliximab Monotherapy in Active Pediatric Crohn's Disease After Immunomodulator Failure
Brief Title: Comparison of 2 Immunomodulator Withdrawal Schemes for Infliximab Monotherapy in Active Pediatric Crohn's Disease After Thiopurine Failure
Acronym: WITHDRAW
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of budget and failure to reach milestones
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0169-12-WOMC
Record Dates: First submitted 2012-12-24; First posted 2013-03-01 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Crohn's Disease
Keywords: Pediatric; Crohn's disease; Infliximab; Thiopurine
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Methotrexate; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunomodulator therapy 26 weeks (Experimental): IFX 5mg/kg for 76 weeks, continuing immunomodulator for 6 months from first infusion
  Interventions: Drug: AZATHIOPRINE or METHOTREXATE
- Immunomodulator therapy 2 weeks (Experimental): IFX 5mg/kg induction for 76 weeks, discontinuing immunomodulator on day of second infusion( after 14 days).
  Interventions: Drug: AZATHIOPRINE or METHOTREXATE

INTERVENTIONS:
Drug: AZATHIOPRINE or METHOTREXATE — Patients should continue azathioprine or 6 MP or methotrexate at their previous doses for 6 months IMM therapy 26 weeks
  Other Names: 6 MERCAPTOPURINE
  Arms: Immunomodulator therapy 26 weeks
Drug: AZATHIOPRINE or METHOTREXATE — Patients should continue the same dose of azathioprine or 6 MP or methotrexate until the day of the second infusion (week 2)
  Thiopurine therapy 2 weeks
  Other Names: 6 MERCAPTOPURINE
  Arms: Immunomodulator therapy 2 weeks

SUMMARY:
The goal of the present study is to evaluate the best regimen for infliximab monotherapy, and to evaluate if limited combination therapy with IFX and an Immunomodulator for the first 6 months of therapy, in prior Immunomodulator failures, is superior to monotherapy with Immunomodulator cessation from the second infusion, in preventing loss of remission to IFX.

DETAILED DESCRIPTION:
Background: Current data from studies and registries involving pediatric Crohn's disease indicate that 50-80% of children will receive an immunomodulator (IMM) as a maintenance therapy within 12 months of diagnosis, and between 60-80% by 18 months. The common use of IMM early in the disease also leads to a high proportion of patients with active disease despite IMM (IMMfailure).

Infliximab has become a standard of care in North America, Europe and Israel, and is recommended at present for steroid dependent or refractory patients, fistulizing disease, active disease despite an immunomodulator.

Infliximab was originally prescribed as an add on therapy to IMM, because of concerns regarding IFX side effects and loss of response due to development of antibodies to infliximab (ATIs). An early study clearly showed an advantage in long term remission with thiopurine co administration.However, subsequent studies in adults with CD showed that with scheduled IFX treatment, AZA could be safely discontinued after the first 6 months of therapy , lowering the risks associated with dual immunosuppressive therapies, and the risks of co-therapy. Monotherapy subsequently became the recommended method of treatment with IFX, despite a decrease in trough levels among those who discontinued IMM.

IFX mono-therapy became the method of choice for treatment in pediatric CD, though this strategy has been called into question due to frequent loss of response to IFX requiring dose escalation of IFX or decreased intervals of IFX. This loss of response has been attributed to development of ATIs and low trough levels of IFX, which can develop after the first infusions. Low trough levels of infliximab at 14 weeks were predictive of LOR. The second reason for questioning IFX mono-therapy is a trial that compared mono-therapy to combined AZA+IFX therapy in adults with moderate to severe thiopurine naïve disease. This study clearly showed improved long term remission rates and mucosal healing in an unselected cohort of patients with combination therapy. Conversely, mono-therapy was associated with low levels of sustained mucosal healing, which is troublesome. Lastly, some excellent results obtained in a pediatric cohort treated with combined therapy, along with the relatively low risk of HTSCL, has left pediatric gastroenterologists at a loss; Should we recommend primary mono-therapy , or use IMM for a limited period of time before discontinuing therapy ? When should the IMM be discontinued, after the first infusion or after several months? There are no controlled data in pediatric IBD to answer this pressing question.

There is also a movement towards increased use of methotrexate instead of thiopurines as immunomodulators because of concerns about neoplasia.

Recent studies have shown that by adding an immunomodulator to a biologic after LOR, trough levels can be improved and ATIs or ADAs decreased, suggesting that IMM may inhibit antibody formation.

The investigators hypothesize that by continuing IMM with IFX for the first 6 months, the investigators will detect a benefit . The investigators hypothesize that early cessation of an IMM will increase the risk of LOR (Loss of response), decrease trough levels at 14 weeks, and be associated with lower rates of corticosteroid free sustained remission by one year.

In a parallel study , using the same data base, We also hypothesize that low trough levels at week 14 ( parallel study) will predict LOR- This study, called Predict Study; Prediction of Loss of Response to Infliximab in Crohn's Disease Based on Week 14 Trough Levels.will enable open label enrolment of patients receiving infliximab with an immunomodulator, but will not require randomization, and patients may be allocated to group one or group 2 at the physicians or patients discretion.

Methods: It is a prospective open label phase 4 RCT in pediatric patients with active CD, defined by the Porto criteria, despite >10 weeks of prior treatment with an immunomodulator (thiopurines/Methotrexate) ,requiring infliximab, involving 2 arms, and intention to treat analysis after the first infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Crohns disease
2. Age: 6 - 18 years ( inclusive)
3. Active disease PCDAI >10, or any steroid dependence despite thiopurine use for >10 weeks.
4. Naïve to biologics
5. Informed consent
6. CRP ≥0.6 mg/dl
7. Neg. TB-Test, negative HBV- S Ag
8. Use of IMM at present or in past for at least 10 weeks ( for Withdraw only).
9. Negative stool culture, parasites and clostridium toxin current flare

Inclusion criteria Comments:

1. Patients receiving corticosteroids may be included if the disease is active and CRP elevated.
2. All other treatments such as 5ASA , , must be discontinued immediately after the first IFX infusion.
3. Patients may receive an antihistamine prior to any infusion.Use of corticosteroid pretreatment is allowed only during the first two infusions (single infusion on day of infliximab), or if an infusion reaction has occurred.
4. Partial enteral nutrition, accounting for less than 50% of daily required calories, may be supplied as needed.
5. Patients receiving antibiotics must cease use of antibiotics within the 14 days of receiving the first infusion.
6. ESR >20 can be alternative if the CRP <0.6.
7. Negative stool culture, parasites and clostridium toxin current flare will examined only if the patient has diarrhea.
8. Patients may be enrolled directly in to the Predict study , in which case duration of IMM is irrelevant , but patients must have received an IMM until week 2 as in the withdraw

Exclusion Criteria:

1. Intolerance to thiopurines/methotrexate
2. Pregnancy
3. Contraindication for any of the drugs.
4. Leukopenia <4000 or absolute neutrophil count below 1200 on two consecutive tests during screening.
5. Hepatocellular Liver disease ( ALT > 60 ) or cirrhosis.
6. Renal Failure
7. Prior idiosyncratic side effects with thiopurines ( pancreatitis etc).
8. Current abscess ( < 14 days of antibiotics) or perforation of the bowel( <14 days antibiotics).
9. Small bowel obstruction within the last 3 months
10. Fixed non inflammatory stricture with predilatation with symptoms related to stricture
11. Complicated or heavily draining perianal fistula ( indolent non draining or scant draining fistula are not exclusion criteria)
12. Prior treatment with infliximab
13. Previous malignancy
14. Toxic Megacolon
15. Sepsis
16. Surgery related to Crohn's disease in previous 8 weeks.
17. Positive Hepatitis B surface antigen or evidence for TB.
18. Current bacterial infection
19. IBD unclassified

Exclusion criteria Comments:

1. Prior surgery or post operative recurrence are not exclusion criteria.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Complete or partial LAR (lack of remission) | 76 weeks
  * Complete LAR- Patient failing to achieve remission after first 3 scheduled doses , or absence of remission 7 days after an infliximab infusion in a patient who had achieved remission after any previous infusion, and unresponsive to dose escalation or dose interval change, or relapse occurring less than 4 weeks after last infusion
  * Partial LAR- Relapse 4-8 weeks after previous infusion, with requirement for dose escalation or shortening of infliximab schedule, and remission with change in dosing or interval.

SECONDARY OUTCOMES:
Mean trough level | 14 and 52 weeks
Sustained steroid free remission | 52 and 76 weeks
Presence of ATI | 52 weeks
Corticosteroid free remission | 14 weeks
Hospitalizations for LOR (loss of response) or failure to obtain remission | Up to 76 weeks
Medication associated adverse events | Up to 76 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Study Chair — Pediatric Gastroenterology and Nutrition Unit, The E. Wolfson MC, Tel-Aviv University, Holon, Israel; Dan Turner, MD, PhD, Study Director — Pediatric Gastroenterology and Nutrition Unit, The Hebrew University of Jerusalem, Shaare Zedek MC, Jerusalem, Israel; Raanan Shamir, MD, Principal Investigator — Schneider Childrens Hospital; Michal Kori, MD, Principal Investigator — Kaplan Medical Center; Michael Wilshanski, MD, Principal Investigator — Hadassah Medical Organization; Ron Shaoul, MD, Principal Investigator — Meyer Childrens Hospital Rambam, Haifa, Israel; Shlomi Cohen, MD, Principal Investigator — Tel Aviv Medical Center; Batia Weiss, MD, Principal Investigator — Sheba Medical Center; Sarit Peleg, MD, Principal Investigator — Afula Hospital; Baruch Yerushalmi, MD, Principal Investigator — Soroka University Medical Center; Efrat Broide, MD, Principal Investigator — Asaf Harofe Medical Center; Avi On, MD, Principal Investigator — Poriah Hospital; Hussein Chemali, MD, Principal Investigator — Nazheret Hospital; Aharon Lerner, MD, Principal Investigator — Carmel Hospital
Locations (1):
- The E. Wolfson.Medical Center, Holon, Israel